CLINICAL TRIAL: NCT02600845
Title: ACCU-CHEK Connect Personal Diabetes Management Study (PDM)
Brief Title: ACCU-CHEK Connect Personal Diabetes Management Study (PDM CONNECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD002206
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ACCU-CHEK (Experimental): All participants will utilize ACCU-CHEK Connect Diabetes Management System containing three primary components: ACCU-CHEK Aviva Connect Blood Glucose Monitoring System intended to be used for the quantitative measurement of glucose, ACCU-CHEK Connect Diabetes Management App indicated as an aid in the treatment of diabetes, and ACCU-CHEK Connect Online Diabetes Management System indicated for use by persons with diabetes or by healthcare professionals in the home or in healthcare facilities.
  Interventions: Device: ACCU-CHEK

INTERVENTIONS:
Device: ACCU-CHEK — ACCU-CHEK Connect Diabetes Management System contains ACCU-CHEK Aviva Connect Blood Glucose Monitoring System, ACCU-CHEK Connect Diabetes Management App, and ACCU-CHEK Connect Online Diabetes Management System.

SUMMARY:
This post-market, interventional, prospective, single arm, the United States (US) based multi-center study will assess the change in treatment satisfaction of participants who utilize the ACCU-CHEK Connect Diabetes Management System over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes for greater than or equal to (>=) 6 months
* Currently using insulin as a component of the diabetes therapy
* Allow and be able to provide self-monitoring of blood glucose (SMBG) data at least 1 month prior to study start
* SMBG frequency as confirmed by site SMBG data download of participants meter(s): Basal insulin treated participants - SMBG >=5 times per week and Multiple dose insulin participants - SMBG >=2 times per day
* Glycosylated hemoglobin (HbA1c) of >=7.5 percentage (per local laboratory obtained less than or equal to [<= 3] months of Baseline)
* Able to read and write in English language
* Currently using a Smartphone and have experience with downloading at minimum one application
* Smartphone compatibility; must be able to download the ACCU-CHEK Connect system application accordingly
* Naive to the ACCU-CHEK Connect system
* Willing to comply with study procedures

Exclusion Criteria:

* Treatment with insulin pump therapy
* Any use of continuous glucose monitoring (CGM) to manage their diabetes during the course of the study
* Visually impaired
* Women who are pregnant, lactating or planning to become pregnant during the study period
* Diagnosed with any clinically significant condition (for example anemia, major organ system disease, infections, psychosis or cognitive impairment)
* Participant requires chronic steroid in adrenal suppressive doses, other immuno-modulatory medication or chemotherapy
* Participant is the investigator or any sub-investigator, general practitioner, practice staff, pharmacist, research assistant or other staff or relative of those directly involved in the conduct of the study and design of the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2017-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lena Borsa, Study Director — Hoffmann-La Roche
Locations (11):
- United States (11):
  - Montgomery, Alabama
  - Huntington Beach, California
  - Atlanta, Georgia
  - Macon, Georgia
  - Ocean Springs, Mississippi
  - Lincoln, Nebraska
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Pottstown, Pennsylvania
  - Bristol, Tennessee
  - Plano, Texas

REFERENCES:
- [Derived] Mora P, Buskirk A, Lyden M, Parkin CG, Borsa L, Petersen B. Use of a Novel, Remotely Connected Diabetes Management System Is Associated with Increased Treatment Satisfaction, Reduced Diabetes Distress, and Improved Glycemic Control in Individuals with Insulin-Treated Diabetes: First Results from the Personal Diabetes Management Study. Diabetes Technol Ther. 2017 Dec;19(12):715-722. doi: 10.1089/dia.2017.0206. Epub 2017 Oct 13. PMID 29027812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified and recruited from the investigators' established subject populations or from the subject populations of other physicians within the group practice, using protocol-specified inclusion and exclusion criteria.
Groups:
- ACCU-CHEK: All participants utilized ACCU-CHEK Connect Diabetes Management System containing three primary components: ACCU-CHEK Aviva Connect Blood Glucose Monitoring System intended to be used for the quantitative measurement of glucose, ACCU-CHEK Connect Diabetes Management App indicated as an aid in the treatment of diabetes, and ACCU-CHEK Connect Online Diabetes Management System indicated for use by persons with diabetes or by healthcare professionals in the home or in healthcare facilities.
Period: Overall Study
Arm/Group | ACCU-CHEK
Started | 122
Completed | 104
Not Completed | 18
Not completed — Reason Not Specified | 3
Not completed — Non-compliance with Study Procedures | 10
Not completed — Consent Withdrawal | 5

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included the full analysis set (FAS), defined as all participants enrolled and trained who had provided data using the ACCU-CHEK Connect system within 14 days of Scheduled Visit 4 during the study, and had completed the Diabetes Treatment Satisfaction Questionnaire (DTSQc) at Week 24.
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction: Diabetes Treatment Satisfaction Questionnaire (DTSQc) Score at Week 24
Description: The Diabetes Treatment Satisfaction Questionnaire for change from Baseline (DTSQc) to study end contains 6 items which can be rated from -3='much worse now' to 3='much better now'). The total score is the sum of the scores of the 6 items and ranges from -18 to 18. A higher score indicates more satisfaction. This questionnaire was administered at the end of the study (Week 24) only.
Time Frame: Week 24
Population: The full analysis set (FAS) was defined as all participants enrolled and trained who had provided data using the ACCU-CHEK Connect system within 14 days of Scheduled Visit 4 during the investigation, and had completed the DTSQc at Week 24.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 87
score on a scale | 14.3 [13.2 to 15.4]

2. Secondary Outcome: Change From Baseline to Week 24 in Diabetes Distress Scale (DDS) Score
Description: Participants rated their level of diabetes distress by answering 17 questions in in the following areas: Regimen-related Distress, Emotional Burden, Diabetes-related Interpersonal Distress and Physician-related Distress (PD) on a 6-point scale: 1=Not a problem to 6=A very serious problem. The Average Total score ranged from 1 (best) to 6 (worst). Results were calculated using a Linear Mixed Model with study group, visit, group-by-visit interaction, baseline DDS, gender, age, and race as fixed effects; and site and subject as random effects. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: The full analysis set (FAS) was defined as all participants enrolled and trained who had provided data using the ACCU-CHEK Connect system within 14 days of Scheduled Visit 4 during the investigation, and had completed the DTSQc at Week 24. Data from evaluable participants are reported.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 80
score on a scale | -0.3 [-0.4 to -0.2]

3. Secondary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Weeks 12 and 24
Description: Assessment of HbA1c is an indicator of long-term control of diabetes.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 85
percent
  Week 12 | -1.07 (1.384)
  Week 24 | -0.95 (1.588)

4. Secondary Outcome: Mean Change From Baseline to Week 24 in Percentage of Glucose Readings in Target Range
Description: Glucose target range was specified as 70-180 milligrams per deciliter (mg/dL).
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 73
percent | 14.74 (34.018)

5. Secondary Outcome: Change From Baseline to Week 24 in Mean Blood Glucose Level
Description: Blood glucose is a type of sugar in blood and is measured to assess a participant's control of diabetes.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 73
milligrams per deciliter | -24.79 (50.813)

6. Secondary Outcome: Change From Baseline to Week 24 in Glycemic Variability
Description: Glycemic variability refers to swings in blood glucose levels. Mean glycemic variability is expressed as a standard deviation of blood glucose data. A negative number indicates a decrease in glucose variability. A positive number indicates and increase in glucose variability.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 73
milligrams per deciliter (mg/dL) | -9.26 (19.244)

7. Secondary Outcome: Incidence of Hypoglycemia
Description: A hypoglycemic reading was defined as a glucose value that fell below the 70 mg/dL level. The incidence of hypoglycemia was defined as the number of hypoglycemic readings in the interval divided by the total number of blood glucose checks in the interval.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hypoglycemic readings
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 87
hypoglycemic readings
  Baseline: number analyzed (Participants) | 73
  Baseline | 1.45 (3.227)
  Week 12 | 1.08 (2.151)
  Week 24 | 1.48 (3.445)

8. Secondary Outcome: Number of Participants With Competency in Self-monitoring of Blood Glucose (SMBG) at Week 24
Description: Competency was defined as appropriate response to high and low glucose values.
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 97
Participants | 1

9. Secondary Outcome: Percent of Follow-Up Visits With Sufficient SMBG Data
Description: Sufficient SMBG data is based on the ability of the healthcare provider to make informed decisions regarding therapy adjustments.
Time Frame: Up to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of follow-up visits
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 86
percentage of follow-up visits | 91.71 (15.281)

10. Secondary Outcome: Change From Baseline in the Number of Blood Glucose Checks at Weeks 12 and 24
Description: An increase in the number of blood glucose checks indicates more glycemic control.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: blood glucose checks
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 73
blood glucose checks
  Week 12 | 16.25 (35.653)
  Week 24 | 9.37 (35.132)

11. Secondary Outcome: Change From Baseline in Mean Daily Self-Monitoring of Blood Glucose (SMBG) Frequency at Weeks 12 and 24
Description: An increase in SMBG frequency indicates more glycemic control. The average number of daily SMBG measurements per interval was calculated based on the total number of blood glucose readings recorded during the study visit interval.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: glucose checks per day
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 73
glucose checks per day
  Week 12 | 0.45 (1.201)
  Week 24 | 0.22 (1.205)

12. Secondary Outcome: Percentage of Blood Glucose Tagged Data
Description: Tagged data specifies the timing of blood glucose recording and includes: fasting, before breakfast, after breakfast, before lunch, after lunch, before dinner, after dinner, and bedtime. The percentage of blood glucose tagged data per interval was calculated as the total number of tagged blood glucose readings during the interval divided by the total number of readings within the interval.
Time Frame: Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | ACCU-CHEK
Number analyzed (Participants) | 87
percentage
  Week 12: number analyzed (Participants) | 80
  Week 12 | 84.24 (24.461)
  Week 24: number analyzed (Participants) | 78
  Week 24 | 86.87 (21.545)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: The Safety Population included all participants.
Arm/Group | ACCU-CHEK
Serious Adverse Events (participants affected / at risk) | 8/122
Other Adverse Events (participants affected / at risk) | 18/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACCU-CHEK (N=122)
Angina pectoris (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Gastrointestinal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arachnoiditis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACCU-CHEK (N=122)
Hypoglycemia (Metabolism and nutrition disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.